CLINICAL TRIAL: NCT07313215
Title: The Efficacy and Complications of Rifampin-combined Antibiotic Therapy for Staphylococcal Periprosthetic Joint Infections（PJI）: A Multicenter, Randomized Controlled Trial
Brief Title: Rifampin-combined Antibiotic Therapy for Staphylococcal PJI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Xinyu Fang, Deputy chief physician, First Affiliated Hospital of Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRCTA, ECFAH of FMU[2024]821-1
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Periprosthetic Joint Infection
Keywords: Periprosthetic Joint Infection; Debride ment, antibiotics, and implant retention; Revision
MeSH Terms: interventions — Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rifampicin combined with antibiotic treatment group (Experimental): In the "rifampicin combined with antibiotic treatment" group, on the basis of conventional antibiotic treatment, rifampicin is taken orally for an additional three months
  Interventions: Drug: Rifampicin (R)
- antibiotic treatment group (Active Comparator): In the "antibiotic treatment" group, conventional antibiotics alone are used for treatment
  Interventions: Drug: Rifampicin (R)

INTERVENTIONS:
Drug: Rifampicin (R) — In the "rifampicin combined with antibiotic treatment" group, on the basis of conventional antibiotic treatment, rifampicin is taken orally for an additional three months. In the "antibiotic treatment" group, conventional antibiotics alone are used for treatment

SUMMARY:
This is a prospective, multicenter, randomized controlled study. Patients were evaluated through inclusion and exclusion criteria. Patients who meet the conditions will sign an informed consent form. After DAIR surgery, they will be treated with intravenous antibiotics for 1-2 weeks and then randomly assigned to one of the following two groups: Antibiotic treatment group: All enrolled patients will be treated with antibiotics (fluoroquinolones or linezolid) for 3 months based on the results of microbial culture and drug sensitivity after surgery. Rifampicin combined with antibiotics treatment group: In addition to the above-mentioned antibiotics, all enrolled patients were treated with rifampicin for 3 months after the operation. The infection control rates of the two groups were judged through at least 2-year follow-up after the operation.The study will follow the Consolidated Standards of Reporting Trials (CONSORT) guidelines for reporting parallel group randomised trials. Ethical approval will be obtained from each institution. Written informed consent will be obtained from all participants to ensure their voluntary participation and understanding of the study.

DETAILED DESCRIPTION:
This study aims to evaluate the efficacy and safety of combined rifampicin for antibiotic treatment in patients with PJI after surgical treatment Sex. The research subjects were PJI patients with staphylococcus as the pathogen. After receiving DAIR treatment, they were screened and enrolled according to strict inclusion and exclusion criteria and randomly assigned to the rifampicin combined with antibiotic treatment group or the conventional antibiotic treatment group only. Then, systematic follow-up was conducted on the patients. Regularly assess its safety indicators such as the recurrence rate of infection, inflammatory indicators, prosthesis function recovery and drug side effects. The data will be entered through a unified recording system and patients who do not meet the research design will be excluded according to the predetermined exit criteria. After the follow-up, the data were summarized and analyzed, with a focus on examining the differences in the efficacy and safety of rifampicin combined therapy in controlling PJI infection. Through this study, we hope to clarify the efficacy and safety of rifampicin combined with antibiotics in PJI treatment, thereby providing a reference basis for the optimization of antibiotic regimens for PJI.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as PJI according to the MSIS criteria

  * The pathogenic bacteria were identified as Staphylococcus through microbial culture and drug sensitivity tests were conducted

    * There are complete clinical data ④ Age under 80 years old, without serious complications or immunosuppressive status ⑤ The patient voluntarily participated in this study and was physically and mentally tolerant of the treatment process and various tests in this study. They have signed the informed consent form and passed the review of the ethics committees of all hospitals participating in this study

Exclusion Criteria:

* Those with chronic inflammation in other parts of the body before the operation

  * Non-staphylococcal infection or mixed infection

    * The patient has other diseases that may affect the outcome, such as immune deficiency or liver and kidney dysfunction ④ Those with an expected lifespan of less than half a year ⑤ The researcher determined that the patient no longer met the criteria of this study due to compliance issues

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-18 (Estimated)

PRIMARY OUTCOMES:
The clearance rate of infection, calculated by the formula | two years postoperatively
  The number of subjects determined to have cleared the infection/the total number of subjects who completed the follow-up. Infection clearance is defined as the patient's (1) complete eradication of infection, wound healing, no fistula, no drainage, no pain, and no recurrence of the same strain of infection. (2) No reoperation intervention due to infection; (3) No deaths caused by PJI-related diseases such as sepsis and necrotizing fasciitis occurred
Adverse events related to PJI | Two years postoperatively

SECONDARY OUTCOMES:
Postoperative functional score | Two years postoperatively
The rate of prosthesis loosening after surgery, the revision rate, and the proportion of prostheses that need to be removed | Two years postoperatively
The incidence of antibiotic complications | Two years postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Wenming Zhang, MD, Study Director — First Affiliated Hospital of Fujian Medical University
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-11-25): https://cdn.clinicaltrials.gov/large-docs/15/NCT07313215/Prot_SAP_000.pdf
  • Informed Consent Form (2025-11-25): https://cdn.clinicaltrials.gov/large-docs/15/NCT07313215/ICF_001.pdf